CLINICAL TRIAL: NCT07291700
Title: A Non-Interventional Study to Investigate the Effectiveness of Hydrotalcite to Relieve Acid-Related Symptoms Due to an Acid Rebound After Discontinuation of a Non/No Longer Indicated Long-Term PPI Therapy.
Brief Title: Study on Hydrotalcite for Relief of Acid Symptoms Due to Acid Rebound After Stopping Long-Term PPI Therapy
Status: Recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22800
Record Dates: First submitted 2025-11-17; First posted 2025-12-18 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Gastroesophageal Reflux
Keywords: Heartburn,; Gastroesophageal Reflux,; Nausea,; Epigastric Pain,; Feeling of Fullness,; Acid-related Symptoms,; Acid Rebound
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn; Nausea | interventions — hydrotalcite

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Talcid (hydrotalcite) 500mg chewable tablet
  Interventions: Drug: Hydrotalcite (Talcid, BAYX002833)

INTERVENTIONS:
Drug: Hydrotalcite (Talcid, BAYX002833) — Talcid Chewable Tablet (500 mg hydrotalcite) taken on-demand for acid-related symptoms.

SUMMARY:
This observational study aims to explore the effectiveness of hydrotalcite, marketed as Talcid, in alleviating acid-related symptoms that occur due to an acid rebound after discontinuing a non-/no-longer-indicated long-term proton pump inhibitor (PPI) therapy. PPIs are commonly prescribed to reduce stomach acid to alleviate symptoms such as heartburn and for the treatment of, for example, duodenal and stomach ulcers. Discontinuation after prolonged use can lead to a rebound effect where dyspeptic complaints such as heartburn occur once the medication is stopped. This study is conducted in Germany and involves adult participants who have stopped using non-/no-longer-indicated PPIs and are experiencing these rebound symptoms.

Hydrotalcite is recommended by physicians as an on-demand treatment for managing acid-related symptoms. The study seeks to gather real-world evidence on its effectiveness, consumer experience, and acceptance to support claims about its use to relieve acid related symptoms due to an acid rebound. Participants will use hydrotalcite as needed (on demand when symptoms occur) over a four-week period, and will record information about symptom relief, the time it takes for relief to occur, and overall satisfaction with the treatment. Additionally, their doctors rate the suitability, tolerability, and effectiveness of the treatment.

The primary objective of the study is to assess the effectiveness of hydrotalcite by the number and percentage of patients not having used PPIs during the study period. Secondary objectives include evaluating relief from specific symptoms (heartburn, reflux, epigastric pain, feeling of fullness, and nausea, as well as improvements in quality of life due to hydrotalcite treatment. The study will also assess participants' satisfaction with hydrotalcite as an on-demand treatment and its suitability for managing these symptoms.

Participants will be adults aged 18 and older who have discontinued a long-term PPI therapy (≥8 weeks) for which there is no current indication according to indication and guidelines and who are experiencing acid rebound symptoms after stopping the PPI therapy. The study will exclude individuals with endoscopically diagnosed gastroesophageal reflux disease (GERD) (LA grade C/ D esophagitis) or those with hydrotalcite contraindications or warnings, such as pregnancy, severe renal impairment, or allergies to its ingredients.

Data will be collected through standardized questionnaires completed by participants after they consent to join the study. The study aims to enroll approximately 167 participants, anticipating a 40% drop-out rate, to ensure around 100 completed questionnaires. Statistical analyses will be exploratory and descriptive, focusing on categorical and continuous variables.

The study is designed to be observational, meaning there will be no direct intervention or randomization of participants. Instead, it will collect primary data directly from participants and investigators across approximately twenty sites in Germany. The results will provide valuable insights into the effectiveness of hydrotalcite in managing acid rebound symptoms and may inform future treatment recommendations for participants discontinuing long-term PPI therapy.

ELIGIBILITY:
Eligibility Criteria:

Adult female or male subjects aged ≥ 18

* Subjects who have discontinued daily PPI therapy (≥ 8 weeks of therapy) for which there is no current indication according to guidelines and approval status, e.g.

  * irritable bowel syndrome
  * subjects who receive Non-Steroidal Anti-Inflammatory drug (NSAID) treatment with no warning signals* regarding ulcers
  * polymedication** with no warning signals* or side effects regarding ulcers
  * unclarified upper abdominal discomfort
  * mild forms of GERD; like Non-Erosive Reflux Disease (NERD), Los Angeles (LA) grade A/B esophagitis
* Suffer from acid-rebound due to a discontinuation of a non/no longer indicated long-term PPI therapy (≥ 8 weeks of therapy)
* No endoscopically diagnosed GERD***
* No indication for a PPI-therapy according to guidelines.

Examples for guideline recommendations for a PPI-therapy:

* moderate - severe forms of reflux esophagitis
* gastric ulcer, duodenal ulcer
* Helicobacter pylori eradication
* moderate/severe forms of GERD - Los Angeles (LA) grade C/D esophagitis
* Zollinger-Ellison-Syndrome

No Talcid® contraindications or warnings as:

* pregnancy and lactation
* severe renal impairment
* hypophosphatemia
* existing myasthenia gravis
* impaired renal function
* Alzheimer's disease or other forms of dementia
* patients under low-phosphate diet
* hypersensitivity to the ingredients of Talcid®

  * Subjects who voluntarily agree to use Talcid® Chewable Tablets for relief of acid-related symptoms due to acid-rebound
  * Decision to initiate on-demand treatment of acid-related symptoms due to acid-rebound with Talcid® was made as per investigator's routine recommendation practice and by the subject
  * Subject purchases Talcid® for her/his own use
  * Signed informed consent
  * No participation in an investigational program with interventions outside of routine clinical practice
  * No contraindications according to the local marketing authorization

    * Warning signals:
  * Age > 60 (with one additional warning signal)
  * Previous history or family history of ulcers
  * Helicobacter pylori positive status ** Polymedication: defined as at least five medicinal products at the same time for a continuous therapy *** Endoscopy: LA grade C/ D esophagitis, Barrett esophagus, peptic stricture; pH- Impedance measurement: acid exposure > 6%

Exclusion Criteria: not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects aged 18 years and older for whom there is not/no longer an indication for a daily PPI therapy according to approval status and guidelines, and who suffer from acid related symptoms due to an acid rebound after discontinuation of a non/no longer indicated long-term PPI-therapy (≥8 weeks).
Sampling Method: Non-Probability Sample
Enrollment: 167 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Number and percentage of subjects successfully discontinued proton pump inhibitor (PPI) therapy defined as no intake of PPI within a period of 4 weeks after start of treatment | 4 weeks
  Number and percentage of subjects successfully discontinued PPI therapy defined as no intake of PPI within a period of 4 weeks after start of hydrotalcite (500 mg Talcid chewable tablets) as on-demand treatment to treat symptoms due to acid-rebound.

SECONDARY OUTCOMES:
Score (5-point rating scale) of overall relief from acid-related symptoms due to an acid rebound when used as an on-demand treatment | Daily during 4-week treatment period
  Overall relief from acid-related symptoms (by subject): Assessed using a 5-point rating scale (1 = Very Poor, 2
  = Poor, 3 = Moderate, 4 = Good, 5 = Very Good) in the evening after Talcid® Chewable tablet intake.
Number and percentage of subjects satisfied with hydrotalcite (Talcid® Chewable Tablets) as an on-demand treatment for treating their acid-related symptoms due to an acid-rebound | once at the end of the 4-week treatment period
  Overall satisfaction assessment (by subject): Assessed at the end of the 4-week on-demand Talcid® Chewable Tablets treatment period using a 7-point rating scale (1 = Strongly Dissatisfied, 2 = Dissatisfied, 3 = Slightly Dissatisfied; 4 = Neither Satisfied nor Dissatisfied, 5 = Slightly Satisfied, 6 = Satisfied, 7= Strongly Satisfied).
Number and percentage of investigators considering hydrotalcite (Talcid® Chewable tablets) being suitable as an on-demand treatment for treating acid-related symptoms due to an acid-rebound | once at final data collection timepoint at the end of the 4-week treatment period
  Suitability assessment (by Investigator): Assessed at the final data collection timepoint using a 5-point rating scale (1 = Not Suitable, 2 = Not Very Suitable, 3 = Neutral, 4 = Suitable, 5 = Very Suitable).
Number and percentage of investigators considering hydrotalcite (Talcid® Chewable tablets) being well tolerated as an on-demand treatment for treating acid-related symptoms due to an acid-rebound | once at final data collection timepoint at the end of the 4-week treatment period
  Tolerability assessment (by Investigator): Assessed at final data collection timepoint using a 5-point rating scale (1 = Very Poor Tolerability, 2 = Poor Tolerability, 3 = Neutral, 4 = Well Tolerated, 5 = Very Well Tolerated).
Number and percentage of investigators considering hydrotalcite (Talcid® Chewable tablets) being effective as an on-demand treatment for treating acid-related symptoms due to an acid-rebound | once at final data collection timepoint at the end of the 4-week treatment period
  Effectiveness assessment (by Investigator): Assessed at the final data collection timepoint using a 5-point rating scale (1 = Not Effective at All, 2 = Not Very Effective, 3 = Neutral, 4 = Effective, 5 = Very Effective).
Scores (5-point rating scale) of relief from heartburn, reflux, epigastric pain, feeling of fullness, and nausea due to an acid-rebound when used as an on-demand treatment (Talcid® Chewable tablets) | Daily during 4-week treatment period
  Specific symptom relief assessments (by subject): Assessment of relief of heartburn, reflux, epigastric pain, feeling of fullness, nausea in the evening after Talcid® Chewable Tablets intake using a 5-point rating scale (1 = Very Poor, 2 = Poor, 3 = Moderate, 4 = Good, 5 = Very Good).
Time to relief of heartburn, reflux, epigastric pain, feeling of fullness, and nausea following intake of hydrotalcite (Talcid® Chewable tablets) when used on-demand | Daily during 4-week treatment period
  Time to relief assessments (by subject): Assessment of time to relief from each of the following symptoms heartburn, reflux, epigastric pain, feeling of fullness, nausea in the evening after Talcid® Chewable Tablets intake using pre-specified time frames (<5, 5- 10, 10-15, 15-30, 30-60, 60-90 and >90 minutes).
Change in scores (5-point rating scale) of quality of life due to hydrotalcite (Talcid® Chewable tablets) on-demand treatment towards baseline | Baseline and at the end of the 4-week treatment
  Quality of Life Assessment (by subject): Assessed at baseline and at the end of the 4-week ondemand Talcid® Chewable Tablets treatment period using a 5-point category scale (1 = Very Poor, 2 = Poor, 3 = Moderate, 4 =Good , 5 = Very Good )

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Bayer Vital GmbH, Leverkusen
  - Bayer Germany, Wuppertal

IPD SHARING:
Plan to Share IPD: No
Currently, there is no established plan for the sharing of Individual Patient Data (IPD) from this study. The availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA 'Principles for responsible clinical trial data sharing.' This pertains to the scope, timepoint, and process of data access.
  As such, Bayer commits to considering requests from qualified researchers for patient- / study-level clinical trial data, and documents from clinical trials involving medicines and indications approved in the US and EU. However, this commitment does not reflect an active IPD sharing plan. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Researchers can use www.vivli.org to request access to IPD and documents from clinical studies to conduct research. Information on Bayer's criteria for listing studies is provided in the member section of the portal.